CLINICAL TRIAL: NCT02250768
Title: Effects of Granulocyte - Macrophage Colony - Stimulating Factor (GM-CSF) Supplementation in Embryo Culture in Patients With Repeated Implantation Failure
Brief Title: Effects of Embryogen in RIF Patients
Acronym: RIF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Dang Quang Vinh, Dr, Vietnam National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGRH-Embryogen
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Infertility
Keywords: GM-CSF, repeated implantation failure
MeSH Terms: conditions — Infertility | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GM-CSF (Experimental): Injected oocytes were cultured in GM-CSF supplemented media until day of transfer
  Interventions: Biological: GM-CSF

INTERVENTIONS:
Biological: GM-CSF — 2ng/ml of GM-CSF supplemented into culture media

SUMMARY:
The purpose of this study was to investigate the potential effects of Granulocyte-Macrophage Stimulating-Colony Factor (GM-CSF) supplementation in embryo culture for patients with repeated implantation failure (RIF)

DETAILED DESCRIPTION:
60 patients with repeated implantation failure were involved.

RIF was defined as patients failed to conceive (beta-hCG < 5 mIU/mL) after at least 03 embryo transfers (fresh and frozen) with 06 top quality embryos or more.

Ovarian stimulation was performed using GnRH antagonist protocol. All matured oocytes were inseminated by ICSI. Injected oocytes were cultured in medium supplemented with 2ng/ml of GM-CSF (Embryogen, Origio) until day of transfer. Embryo evaluation was performed at ﬁxed time points of 18 and 44 hour after fertilization. Embryo transfer was performed 2 days after ovum retrieval.

Luteal-phase support was provided using progesterone gel (Crinone 8% 90 mg, twice a day; Merck Serono) and estradiol per os (Valiera 2mg, twice a day; Laboratorios Recalcine). Serum hCG was measured 16 days after oocyte retrieval, and if positive, an ultrasound scan was performed at gestational weeks 7 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Normal ovarian reserve (AMH > 1.1 ng/ml)
* Regular menstrual cycle (25 - 34 days)
* Clear informations about at least 3 latest IVF/ET
* Fresh embryo transfer in this cycle
* Endometrial thickness of 10 mm or more

Exclusion Criteria:

* Undergo oocyte donation or in vitro maturation (IVM) cycles
* Using frozen or surgically retrieved sperm
* Adenomyosis, Uterine anomaly, uterine fibroid, hydrosalpinges
* In participation in other studies/interventions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 12 week of gestation

SECONDARY OUTCOMES:
Implantation rate | 7 week of gestation
clinical pregnancy rate | 7 week of gestation
top quality embryo rate | 44 hours after insemination

CONTACTS AND LOCATIONS:
Overall Officials: Vinh Q Dang, Dr, Principal Investigator — Research Center for Genetics and Reproductive Health
Locations (2):
- Vietnam (2):
  - An Sinh Hospital, Ho Chi Minh City, Ho Chi Minh
  - An Sinh Hospital, Ho Chi Minh City